CLINICAL TRIAL: NCT05663671
Title: Evaluate Established Anti-DEFA5 mAbs Diagnostic Efficacy and Safety in IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meharry Medical College (Other)
Responsible Party: Principal Investigator, Amosy M'Koma, Professor, Meharry Medical College
Other Study IDs: 22-08-1235
Record Dates: First submitted 2022-11-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Colitis; Indeterminate Colitis
Keywords: Inflammatory bowel disease; Crohn's colitis; Ulcerative colitis; Indeterminate colitis; DEFA5; Molecular diagnostics; Colonic biopsies
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The research outlined is consistent with the Non-human Welfare Act Criteria because investigators receive de-identified specimens and data from an IRB approved repository, and investigators do not have access to the link by which investigators may re-identify the specimens and data with their source. The research involves the use of human tissue acquired previously using the third-party good faith broker mechanism. Since all identifiers are striped, the tissue samples are considered non-human subjects. Each specimen is assigned a unique barcode identifier to maintain the patient's confidentiality. In no case is the patient's name ever revealed to the users. All information accompanying the specimen(s) uses the bar code identifier.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Crohn's colitis: Correlate patient longitudinal study of clinical data and their biopsy data. Investigators will determine DEFA5 levels from endoscopy biopsies from known authentic CC patients.
  Interventions: Diagnostic Test: Diagnostic Test
- Ulcerative colitis: Correlate patient longitudinal study of clinical data and their biopsy data. Investigators will determine DEFA5 levels from endoscopy biopsies from known authentic UC patients.
  Interventions: Diagnostic Test: Diagnostic Test
- Indeterminate colitis: Correlate patient longitudinal study of clinical data and their biopsy data. Investigators will determine DEFA5 levels from endoscopy biopsies from known IC patients (into authentic UC and CC)
  Interventions: Diagnostic Test: Diagnostic Test
- Diverticulitis: Correlate patient longitudinal study of clinical data and their biopsy data. Investigators will determine DEFA5 levels from endoscopy biopsies from known diverticulitis.
  Interventions: Diagnostic Test: Diagnostic Test
- Ileum: Positive control
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — 30% of IBD patients are misdiagnosed. This affects surgical care of patients. Investigators have unveiled a signature discriminator between UC&CC that also predicts the outcome of IC patients into authentic UC/CC. This is a bioassay that is specific, sensitive, linear, affordable, minimal risk, non-invasive and constitutes an inexpensive, simple to use, point-of-care test format. Investigators published data which have shown robust presence of DEFA5 in the colon crypt mucosa with aberrant expression of apparent crypt-cell-like cells (CCLCs) in areas identified with ectopic colon ileal metaplasia consistent with CC. Investigators propose to validate that UC/CC, the two unsolved medical sub-types of pathology can accurately be distinguished among IC patients by examining CCLCs secreted DEFA5 levels in endoscopy biopsies instantly. Diagnostics relies on the expression/localization/activation of DEFA5 and the ectopic CCLCs in the mucosal crypt of CC patients.

SUMMARY:
Investigators propose to validate efficacy and safety of the detection of DEFA5 in the diagnosis of the colonic IBD using longitudinal vs. cross-sectional studies of known patient clinical data to correlate with their endoscopy biopsy data. 30% of colonic IBD patients cannot be accurately diagnosed (CC vs. UC) in a timely manner even when a state-of-the-art classification system of combined clinical, endoscopic, radiologic and histologic tools are used. When the diagnostic classification for these two diseases is inconclusive, the condition is termed indeterminate colitis (IC). Here, the central medical challenge is the discrimination of IBD into the specific subtypes with high accuracy, as it greatly effects surgical care of patients. Diagnostic accuracy of IC into either authentic UC or CC is of utmost importance when determining a patient's candidacy for RPC-IPAA surgery, the standard curative surgical procedure for UC. Further, incorrect diagnosis and treatment carry potential morbidity from inappropriate and unnecessary surgery and costs. The success outcomes of RPC-IPAA surgery and convalescence depend on correct diagnosis. To address IBD diagnosis ambiguity and delays in IBD clinical settings, investigators developed a proteomic signature to discriminate between UC and CC patients that also will predict the outcome of IC patients for their eventual progress to either UC or CC. Our published data has shown robust evidence supporting presence of human alpha-defensin 5 (DEFA5) in areas of the colon mucosa with aberrant expression of apparent Paneth cell-like cells (PCLCs) or crypt cell-like cells (CCLCs), which identifies an area of colonic ileal metaplasia, consistent with the diagnosis of CC. DEFA5 bioassay discriminated CC and UC in a cohort of all IC patients with accuracy. A fit logistic model with group CC and UC as the outcome and the DEFA5 as independent variable differentiator with a positive predictive value of 96%. These findings were obtained solely from colectomy specimens for both the discovery and validation analyses. Investigators believe that use of endoscopy biopsies would be indifferent, which is the purpose of this prospective patient centered clinical study. Investigators propose to demonstrate that UC and CC, the two unsolved medical subtypes of pathology with no drugs for a cure, can accurately be distinguished molecularly by examining CCLCs-secreted DEFA5 in colonic endoscopy biopsies instantly. Our proposal is highly innovative, as it highlights the robustness of DEFA5 and its clinical relevance to IBD is both in science and the anticipated impact, as investigators seek to better understand difficulty to determine 'subtypes" and translate that to improve diagnosis, treatment, clinical outcomes, and quality of life for patients and the realm of clinical care. DEFA5 immunoreactivity in colonic endoscopy biopsies could be a rapid potential diagnostic signature to resolve IC into authentic UC and CC with a first clinic endoscopy biopsy. IC is likely to be eliminated for good.

DETAILED DESCRIPTION:
The clinical relevance of this proposed screen is that it would lead to the elusive and accurate diagnosis to circumvent the inexact IC patients into authentic CC and UC with a first clinic endoscopy biopsy. The central medical challenge in endoscopic medicine and colorectal surgery is the discrimination of colonic IBD into the subtypes with high accuracy because it greatly affects surgical care of patients. Incorrect diagnosis and surgery carry potential morbidity from inappropriate and unnecessary surgery and cost. Our published data has shown robust evidence supporting presence of human alpha-defensin 5 (DEFA5) in areas of the colon mucosa with aberrant expression of apparent Paneth cell-like cells (PCLCs) / crypt cell-like cells (CCLCs), which identifies an area of colonic ileal metaplasia, consistent with the diagnosis of CC. Investigators propose to demonstrate that UC and CC, the two unsolved medical subtypes of GI pathology with no drugs for a cure, may accurately be distinguished molecularly by examining CCLCs-secreted DEFA5 in colonic endoscopy biopsies instantly. Our proposal is highly innovative, as it highlights the robustness efficacy and safety of DEFA5 and its clinical relevance in IBD diagnostics. The goal of this proposal is to develop a clinical approach to circumvent diagnostic ambiguity and delay, as well as permit timely, and accurate diagnosis of colonic IBD. DEFA5 immunoreactivity in colonic endoscopy biopsies could be a potential diagnostic signature that accurately diagnoses CC and provides the basis to resolve ambiguity in the diagnosis of IBD to not only circumvent diagnostic delay, but also permit timely, accurate diagnosis and timely prescription of appropriate treatment options, an Affordable, Sensitive, Specific, User-friendly, Robust and Rapid, Equipment-free, and Deliverable (ASSURED) bioassay that may delineate subtypes of IBD during the first clinic endoscopy biopsy visit. This bioassay is specific, sensitive, linear, affordable, low risk, and less invasive. Investigators hypothesize that aberrant expression of DEFA5 secreting CCLCs in colonic crypt of IBD patients may be exploited as a reliable diagnostic signature to highly differentiate CC from UC in otherwise IC patients during the first clinic visit endoscopy biopsy without delay. Investigators foresee no issues pertaining to this proposal as an established sampling error by endoscopic biopsy making it does not interfere with results and apropos of this project that each biopsy has complement CCLCs with co-localized DEFA5 clearly restricted in areas of the mucosa with aberrant CCLCs identifies a ubiquitously colonic ileal metaplasia that is consistent with the diagnosis of authentic CC. If successful, widespread use of this approach would not only revolutionize provide accurate diagnoses and the correct treatment regimens for IBD patients, but also it will improve health outcomes and patient quality of life, while reducing medical complications and/or unnecessary drugs, surgeries, & costs.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of COLONIC inflammatory bowel disease (IBD) and non-IBD

* COLONIC IBD

  * Colonic Crohn's disease (Crohn's colitis)
  * Ulcerative colitis
  * Indeterminate colitis
* COLONIC non-IBD

  * Diverticulosis
* CONTROL

  * Ileum (positive control)

Exclusion Criteria:

* Patients with IBD under prescription
* Patients with non-colonic IBD
* Children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Using the result of our pilot study of DEFA5 biomarker statistical power analysis, a sample size of 230 subjects is sufficient to detect a clinically significant difference of 19% between the PPVs of CC and UC using a one-tailed test of proportions between the two groups with 80% statistical power and a 5% level of significance. This 19% difference represents 80% probability that subjects in the CC group with a positive screening test truly have the disease and 77% PPV for subjects in UC group. We decided to add non-IBD samples, 46 in the DV arm and 46 in CP arm to strengthen the results.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate Established Anti-DEFA5 mAbs Diagnostic Efficacy and Safety in IBD | Six moths
  Using Western blot (WB) technology investigators will evaluate our newly established Anti-DEFA5 mAbs by measuring and quantifying DEFA5 protein levels in colonic biopsies from IBD and non-IBD patients. Anti-DEFA5 monoclonal antibodies (mAbs), i.e., clones 1A8 & 4FD efficacy. Anti-DEFA5 mAbs specificity and sensitivity to the DEFA5 protein which is diagnostic for colonic Crohn's disease

SECONDARY OUTCOMES:
Evaluate Established Anti-DEFA5 mAbs Diagnostic Efficacy and Safety in IBD | Six months
  Our two newly developed mAbs will be tested by measuring detection sensitivity specific to peptide DEFA5 protein. DEFA5 detection level between the mAbs will determine the most effective Anti-DEFA5 mAb to be used to develop bioassay kit for DEFA5.
Evaluate Established Anti-DEFA5 mAbs Diagnostic Efficacy and Safety in IBD | 12 months
  Using immunohistochemistry (IHC) technology investigators will evaluate diagnostic efficacy and safety of DEFA5 bioassay using colonic IBD biopsies. The DEFA5 protein, which is diagnostic in IBD will be measured and quantified in the colonic biopsies. Investigators will use colon tissue biopsies from patients with UC, CC, IC, diverticulitis, normal (diverticilosis),& ileum as positive control and compare between different pathologies.

CONTACTS AND LOCATIONS:
Overall Officials: Amosy E M'Koma, MD, MS, PhD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be obtained (i) directly with study PI or (ii) request via a data repository

REFERENCES:
- [Result] Williams AD, Korolkova OY, Sakwe AM, Geiger TM, James SD, Muldoon RL, Herline AJ, Goodwin JS, Izban MG, Washington MK, Smoot DT, Ballard BR, Gazouli M, M'Koma AE. Human alpha defensin 5 is a candidate biomarker to delineate inflammatory bowel disease. PLoS One. 2017 Aug 17;12(8):e0179710. doi: 10.1371/journal.pone.0179710. eCollection 2017. PMID 28817680
- [Result] Rana T, Korolkova OY, Rachakonda G, Williams AD, Hawkins AT, James SD, Sakwe AM, Hui N, Wang L, Yu C, Goodwin JS, Izban MG, Offodile RS, Washington MK, Ballard BR, Smoot DT, Shi XZ, Forbes DS, Shanker A, M'Koma AE. Linking bacterial enterotoxins and alpha defensin 5 expansion in the Crohn's colitis: A new insight into the etiopathogenetic and differentiation triggers driving colonic inflammatory bowel disease. PLoS One. 2021 Mar 9;16(3):e0246393. doi: 10.1371/journal.pone.0246393. eCollection 2021. PMID 33690604
- [Result] Ballard BR, M'Koma AE. Gastrointestinal endoscopy biopsy derived proteomic patterns predict indeterminate colitis into ulcerative colitis and Crohn's colitis. World J Gastrointest Endosc. 2015 Jun 25;7(7):670-4. doi: 10.4253/wjge.v7.i7.670. PMID 26140094
- [Result] Korolkova OY, Myers JN, Pellom ST, Wang L, M'Koma AE. Characterization of Serum Cytokine Profile in Predominantly Colonic Inflammatory Bowel Disease to Delineate Ulcerative and Crohn's Colitides. Clin Med Insights Gastroenterol. 2015 May 6;8:29-44. doi: 10.4137/CGast.S20612. eCollection 2015. PMID 26078592
- [Result] M'Koma AE. Diagnosis of inflammatory bowel disease: Potential role of molecular biometrics. World J Gastrointest Surg. 2014 Nov 27;6(11):208-19. doi: 10.4240/wjgs.v6.i11.208. PMID 25429322
- [Result] Seeley EH, Washington MK, Caprioli RM, M'Koma AE. Proteomic patterns of colonic mucosal tissues delineate Crohn's colitis and ulcerative colitis. Proteomics Clin Appl. 2013 Aug;7(7-8):541-9. doi: 10.1002/prca.201200107. Epub 2013 May 8. PMID 23382084
- [Result] M'Koma AE, Seeley EH, Washington MK, Schwartz DA, Muldoon RL, Herline AJ, Wise PE, Caprioli RM. Proteomic profiling of mucosal and submucosal colonic tissues yields protein signatures that differentiate the inflammatory colitides. Inflamm Bowel Dis. 2011 Apr;17(4):875-83. doi: 10.1002/ibd.21442. Epub 2010 Aug 30. PMID 20806340

DOCUMENTS (1):
  • Study Protocol (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT05663671/Prot_000.pdf